CLINICAL TRIAL: NCT02772133
Title: Circulating PRCP in STEMI Patients Undergoing Primary PCI
Status: Completed | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Pan-Pan Hao, MD, PhD, Qilu Hospital of Shandong University
Other Study IDs: 2015GSF118133
Record Dates: First submitted 2016-05-09; First posted 2016-05-13 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Myocardial Infarction; Percutaneous Coronary Intervention; PRCP
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- STEMI patients
  Interventions: Procedure: Primary PCI
- Healthy subjects
- Unstable angina

INTERVENTIONS:
Procedure: Primary PCI
  Groups: STEMI patients

SUMMARY:
Purpose: The purpose of this study is to evaluate the impact of acute ST-segment elevation myocardial infarction (STEMI) and primary percutaneous coronary intervention (PCI) on circulating prolylcarboxypeptidase (PRCP) level and activity.

ELIGIBILITY:
Inclusion Criteria:

* Admitted for primary PCI for STEMI involving the LAD within 12 hours of onset of symptoms. STEMI will be defined as typical ECG changes (ST segment elevation ≥2mm in 2 or more precordial leads) associated with acute chest pain or an elevation of cardiac enzymes;
* Age ≥18 years;
* Informed consent from subject or next of kin.

Exclusion Criteria:

* Nonischaemic Cardiomyopathy;
* Cardiac surgery planed in the 6 months;
* Mechanical complication of STEMI (ventricular septal rupture, free wall rupture, acute severe mitral regurgitation);
* Renal or hepatic failure;
* Malignancy, HIV, or central nervous system disorder;
* Cardiopulmonary resuscitation >15 min and compromised level of consciousness;
* Cardiogenic shock;
* Current participation in any research study involving investigational drugs or devices;
* No written consensus;
* Previous myocardial infarction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects, consecutive patients with unstable angina, and those undergoing primary PCI for STEMI
Sampling Method: Non-Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2016-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Circulating PRCP level | 1 month
Circulating PRCP activity | 1 month

SECONDARY OUTCOMES:
Circulating Ang II level | 1 month
Circulating Ang-(1-7) level | 1 month
Circulating BK-(1-9) level | 1 month
Circulating KBK-(1-9) level | 1 month

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Qianfoshan Hospital, Shandong University, Jinan, Shandong
  - Shandong University Qilu Hospital, Jinan, Shandong
  - Jinan Central Hospital, Shandong University, Jinan, Shandong
  - Shandong Provincial Hospital, Shandong University, Jinan, Shandong